CLINICAL TRIAL: NCT06175702
Title: Treatment Protocol for Newky Diagnosed Adult Ph-Chromosome Positive (BCR::ABL1) Acute Lymphoblastic Leukemia (LALPh2022)
Brief Title: Treatment Protocol for Newky Diagnosed Adult Ph Positive ALL
Acronym: LALPh2022
Status: Not yet recruiting | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PETHEMA LALPh2022
Record Dates: First submitted 2023-11-17; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Lymphoblastic Leukemia; Philadelphia-Positive ALL; Adult ALL
Keywords: Acute Lymphoblastic Leukemia; Philadelphia (BCR::ABL1) positive; Adults
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Dexamethasone; Imatinib Mesylate; Cytarabine; Mercaptopurine; Methotrexate; ponatinib; Whole-Body Irradiation; Cyclophosphamide; fludarabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complete molecular response and low risk genetics: Patients in Complete Remission and Complete Molecular Response at end Induction therapy will receive consolidation with imatinib (or dasatinib if intolerance) and chemotherapy, unless they show the IKZF1plus genotype, which will imply switch to the not complete molecular response or high-risk genetics (IKZ1plus) group.
  Interventions: Drug: Vincristine; Drug: Dexamethasone; Drug: Imatinib; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Methotrexate
- Not complete molecular response or high-risk genetics (IKZF1plus): Patients in Complete Remission and without Complete Molecular Response at the end of Induction therapy or showing the IKZF1plus genotype, will receive consolidation treatment with ponatinib and chemotherapy followed by allogeneic stem cell transplantation and maintenance therapy.
  Interventions: Drug: Vincristine; Drug: Dexamethasone; Drug: Imatinib; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Ponatinib; Procedure: allogeneic stem cell transplantation; Procedure: Total body irradiation; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Vincristine — dose 1.5 mg/m2 at days 1, 8, 15 and 22
Drug: Dexamethasone — 40 mg on days 1-2, 8-9,15-16 and 22-23
Drug: Imatinib — 600 mg per day from 1 to up to 5 years
Drug: Cytarabine — 1000 mg/m2/ on days 1, 3 and 5 of consolidation with 2h infusion
Drug: Mercaptopurine — 50 mg/m2 on days 1 to 28 of maintenance
Drug: Methotrexate — 1000 mg/m2 on day 1 of consolidation with 24h infusion; and 20 mg/m2 on days 1, 8, 15 and 22 of maintenance
Drug: Ponatinib — 15 mg per day from consolidation start up to 5 years
  Groups: Not complete molecular response or high-risk genetics (IKZF1plus)
Procedure: allogeneic stem cell transplantation — Allogeneic stem cell transplantation from hematpoietic stem cells progenitors of familiar or not familiar origin. Cord blood transplantation can also be done.
  Groups: Not complete molecular response or high-risk genetics (IKZF1plus)
Procedure: Total body irradiation — Fractionated dose with total dose of 12 Gy between days -4 and -1 of allogeneic stem cell transplantation (alloSCT)
  Groups: Not complete molecular response or high-risk genetics (IKZF1plus)
Drug: Cyclophosphamide — 60 mg/kg on days -6 and -5 before alloSCT
  Groups: Not complete molecular response or high-risk genetics (IKZF1plus)
Drug: Fludarabine — 30 mg/m2 intravenous on days -7, -6, -5 y -4 before alloSCT (alternative to cyclophosphamide)
  Groups: Not complete molecular response or high-risk genetics (IKZF1plus)

SUMMARY:
The goal of this prospective, multicenter, open observational study is to assess the efficacy and safety of the treatment for acute lymphoblastic leukemia Ph' positive adult patients with approved combinations of chemotherapy and tyrosine kinase inhibitor (TKI).

Efficay refers to the rate of Complete Molecular Response (BCR::ABL1/ABL1 ratio 0.01%) in eah treatment arm. Safety refers to measurement of i) Adverse events (AEs) and serious adverse events (SAEs) according to standard clinical and laboratory tests (hematology and chemistry, physical examination, vital sign measurements, and diagnostic tests), ii) incidence and degree of cytopenias and iii) incidence and degree of infections.

Low-dose chemotherapy will be given together with the TKI imatinib to patients of all ages as induction to remission phase.

Consolidation treatment will continue with low-dose chemotherapy with imatinib if the patient fullfills both criteria: to show a measurable residual disease (MRD) value lower than 0,01% at 3 month of therapy, and not showing IKZF1plus genetics Those patients have any of these 2 conditions will be considered high-risk patients and will recieve consolidation treatment intensification with low-dose chemotherapy plus ponatinib as TKI and allogeneic stem cell transplantation (allo SCT). The remaining patients (standard-risk) will receive maintenance chemotherapy together with imatinib or ponatinib and will not be submitted to alloSCT.

DETAILED DESCRIPTION:
The goal of this prospective, multicenter, open observational study is to assess the efficacy and safety of the treatment for acute lymphoblastic leukemia Ph' positive adult patients with approved combinations of chemotherapy and tyrosine kinase inhibitor (TKI).

Efficay refers to the rate of Complete Molecular Response (BCR::ABL1/ABL1 ratio 0.01%) in each treatment arm. Safety refers to measurement of i) Adverse events (AEs) and serious adverse events (SAEs) according to standard clinical and laboratory tests (hematology and chemistry, physical examination, vital sign measurements, and diagnostic tests), ii) incidence and degree of cytopenias and iii) incidence and degree of infections.

Low-dose chemotherapy induction phase with vincristine (dose 1.5 mg/m2 at days 1, 8, 15 and 22), dexamethasone (dose 40 mg days 1-2, 8-9,15-16 and 22-23) will be given together with the TKI imatinib (dose 600 mg from day to consolidation start) to all patients of all ages as induction to remission phase.

Consolidation treatment will continue with low-dose chemotherapy with methotrexate (dose 1000 mg/m2 on day 1 with 24h infusion) and arabinoside of cytarabine (dose 1000 mg/m2/ days 1, 3 and 5 with 2h infusion) with imatinib (dose 600 mg per day) if the patient fullfills both criteria: i) to show a measurable residual disease (MRD) value <0,01% at 3 month of therapy, and ii) not showing IKZF1plus genetics.

Those patients having any of these 2 conditions will be considered high-risk patients and will recieve consolidation treatment intensification with low-dose chemotherapy (same as described above) plus ponatinib (dose 30 mg per day) as TKI and allogeneic stem cell transplantation (alloSCT) followed by maintenance chemotherapy with mercaptopurine (dose 50 mg/m2 on days 1 to 28) and methotrexate (dose 20 mg/m2 on days 1, 8, 15 and 22) together with imatinib (dose 600 mg per day) or ponatinib (15 mg per day) up to 5 years. The remaining patients (standard-risk) will receive maintenance chemotherapy (as described above) together with imatinib (dose 600 mg per day) or ponatinib (15 mg per day) up to 5 years and will not be submitted to alloSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with de novo avute lymphoblastic leukeima (ALL) Philadelphia chromosome-positive (BCR::ABL1) aged ≥18 years.
2. CML blast crisis will be included. These patients will always receive transplantation, regardless of the molecular response or the genetic risk, following the recommendations of the SEHH CML group (Chronic Myleoid Leukemia Group from the Spanish Society of Hematology).
3. Performance status 0-2; patients with performance status>2 attributable to ALL can be included.
4. Patients without functional alteration of organs; liver function: total bilirubin, GOT, GPT, GGT and alkaline phosphatase less than 3 times the upper limit of the normal range of the laboratory; renal function: serum creatinine <2 mg/dl or creatinine clearance > 30 ml/min (except altered renal function attributable to ALL); normal heart function: EF ventricular > 50%; absence of severe chronic respiratory disease. In case that the alterations are secondary to the disease, it is at the discretion of the physician to determine if the patient can be included in the study.

Exclusion Criteria:

1. Any other subtype of ALL.
2. Patients with chronic liver disease.
3. Patients with chronic respiratory failure.
4. Renal failure not due to ALL.
5. Lipase and amylase>1.5× ULN.
6. Patients with positive HIV serology.
7. Serious neurological alterations not due to ALL.
8. Serious general condition condition (grades 3 or 4 on the WHO scale) not attributable to ALL.
9. Pregnant or breastfeeding women.
10. Impaired cardiac function (defined by an ejection fraction less than 50%), any clinically significant active or uncontrolled cardiovascular condition, uncontrolled hypertension, arrhythmias, ischemic cardiovascular or neurological events, deep vein thrombosis, pulmonary thromboembolism, history of acute pancreatitis in the year before diagnosis of ALL or history of chronic pancreatitis and triglycerides >450 mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 or over years with newly diagnosed Ph-positive or BCR::ABL1-positive acute lymphoblastic leukemia (Ph+ ALL).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-25 (Estimated); Primary Completion 2028-12-25 (Estimated); Study Completion 2030-12-25 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 Years
  Improvement of OS compared to that observed in the previous protocols (PETHEMA LALPh08 and LALOPh07).

SECONDARY OUTCOMES:
Change the complete molecular response (CMR) rate with Ponatinib | 5 Years
  Change the CMR rate at the end of consolidation with the administration of ponatinib to those patients who do not achieve CMR at the end of induction or have high-risk genetics (IKZF1plus).
Limit the number of alloTPH compared to that observed in the previous protocols (PETHEMA LALPh08 and LALOPh07). | 5 Years
  Limit the number of alloTPH to any of the following:
  * Lack of CMR at the end of consolidation.
  * High-risk genetics (IKZF1plus).
Maintenance | 5 Years
  To assess the number of non-transplanted participants who receive maintenance treatment.
Treatment with TKI after HSCT | 5 Years
  To assess the number of transplanted patients who receive TKI maintenance treatment preemptively (upon of MRD>0.01%).
Assess the frequency and degree of Adverse Events | 5 Years
  Assess the frequency of cytopenias and degree. Assess the frequency of infections and degree. Assess the frequency of vascuar events and degree. Assess the frequency of hepatic events and degree. Assess the frequency of pancreatic events and degree.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Ribera Santasusana, MD, Principal Investigator — Institut Catala d'Oncologia-Hospital Universitari Germans Trias i Pujol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiaretti S, Vitale A, Cazzaniga G, Orlando SM, Silvestri D, Fazi P, Valsecchi MG, Elia L, Testi AM, Mancini F, Conter V, te Kronnie G, Ferrara F, Di Raimondo F, Tedeschi A, Fioritoni G, Fabbiano F, Meloni G, Specchia G, Pizzolo G, Mandelli F, Guarini A, Basso G, Biondi A, Foa R. Clinico-biological features of 5202 patients with acute lymphoblastic leukemia enrolled in the Italian AIEOP and GIMEMA protocols and stratified in age cohorts. Haematologica. 2013 Nov;98(11):1702-10. doi: 10.3324/haematol.2012.080432. Epub 2013 May 28. PMID 23716539
- [Background] Fielding AK, Rowe JM, Buck G, Foroni L, Gerrard G, Litzow MR, Lazarus H, Luger SM, Marks DI, McMillan AK, Moorman AV, Patel B, Paietta E, Tallman MS, Goldstone AH. UKALLXII/ECOG2993: addition of imatinib to a standard treatment regimen enhances long-term outcomes in Philadelphia positive acute lymphoblastic leukemia. Blood. 2014 Feb 6;123(6):843-50. doi: 10.1182/blood-2013-09-529008. Epub 2013 Nov 25. PMID 24277073
- [Background] Ribera JM, Oriol A, Gonzalez M, Vidriales B, Brunet S, Esteve J, Del Potro E, Rivas C, Moreno MJ, Tormo M, Martin-Reina V, Sarra J, Parody R, de Oteyza JP, Bureo E, Bernal MT; Programa Espanol de Tratamiento en Hematologia; Grupo Espanol de Trasplante Hemopoyetico Groups. Concurrent intensive chemotherapy and imatinib before and after stem cell transplantation in newly diagnosed Philadelphia chromosome-positive acute lymphoblastic leukemia. Final results of the CSTIBES02 trial. Haematologica. 2010 Jan;95(1):87-95. doi: 10.3324/haematol.2009.011221. Epub 2009 Oct 1. PMID 19797728
- [Background] Daver N, Thomas D, Ravandi F, Cortes J, Garris R, Jabbour E, Garcia-Manero G, Borthakur G, Kadia T, Rytting M, Konopleva M, Kantarjian H, O'Brien S. Final report of a phase II study of imatinib mesylate with hyper-CVAD for the front-line treatment of adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Haematologica. 2015 May;100(5):653-61. doi: 10.3324/haematol.2014.118588. Epub 2015 Feb 14. PMID 25682595
- [Background] Chiaretti S, Vitale A, Vignetti M, Piciocchi A, Fazi P, Elia L, Falini B, Ronco F, Ferrara F, De Fabritiis P, Luppi M, La Nasa G, Tedeschi A, Califano C, Fanin R, Dore F, Mandelli F, Meloni G, Foa R. A sequential approach with imatinib, chemotherapy and transplant for adult Ph+ acute lymphoblastic leukemia: final results of the GIMEMA LAL 0904 study. Haematologica. 2016 Dec;101(12):1544-1552. doi: 10.3324/haematol.2016.144535. Epub 2016 Aug 11. PMID 27515250
- [Background] Chalandon Y, Thomas X, Hayette S, Cayuela JM, Abbal C, Huguet F, Raffoux E, Leguay T, Rousselot P, Lepretre S, Escoffre-Barbe M, Maury S, Berthon C, Tavernier E, Lambert JF, Lafage-Pochitaloff M, Lheritier V, Chevret S, Ifrah N, Dombret H; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL). Randomized study of reduced-intensity chemotherapy combined with imatinib in adults with Ph-positive acute lymphoblastic leukemia. Blood. 2015 Jun 11;125(24):3711-9. doi: 10.1182/blood-2015-02-627935. Epub 2015 Apr 15. PMID 25878120
- [Background] Foa R, Vitale A, Vignetti M, Meloni G, Guarini A, De Propris MS, Elia L, Paoloni F, Fazi P, Cimino G, Nobile F, Ferrara F, Castagnola C, Sica S, Leoni P, Zuffa E, Fozza C, Luppi M, Candoni A, Iacobucci I, Soverini S, Mandelli F, Martinelli G, Baccarani M; GIMEMA Acute Leukemia Working Party. Dasatinib as first-line treatment for adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Blood. 2011 Dec 15;118(25):6521-8. doi: 10.1182/blood-2011-05-351403. Epub 2011 Sep 19. PMID 21931113
- [Background] Ravandi F, Othus M, O'Brien SM, Forman SJ, Ha CS, Wong JYC, Tallman MS, Paietta E, Racevskis J, Uy GL, Horowitz M, Takebe N, Little R, Borate U, Kebriaei P, Kingsbury L, Kantarjian HM, Radich JP, Erba HP, Appelbaum FR. US Intergroup Study of Chemotherapy Plus Dasatinib and Allogeneic Stem Cell Transplant in Philadelphia Chromosome Positive ALL. Blood Adv. 2016 Dec 27;1(3):250-259. doi: 10.1182/bloodadvances.2016001495. PMID 29046900
- [Background] Sugiura I, Doki N, Hata T, Cho R, Ito T, Suehiro Y, Tanaka M, Kako S, Matsuda M, Yokoyama H, Ishikawa Y, Taniguchi Y, Hagihara M, Ozawa Y, Ueda Y, Hirano D, Sakura T, Tsuji M, Kamae T, Fujita H, Hiramoto N, Onoda M, Fujisawa S, Hatta Y, Dobashi N, Nishiwaki S, Atsuta Y, Kobayashi Y, Hayakawa F, Ohtake S, Naoe T, Miyazaki Y. Dasatinib-based 2-step induction for adults with Philadelphia chromosome-positive acute lymphoblastic leukemia. Blood Adv. 2022 Jan 25;6(2):624-636. doi: 10.1182/bloodadvances.2021004607. PMID 34516628
- [Background] Kim DY, Joo YD, Lim SN, Kim SD, Lee JH, Lee JH, Kim DH, Kim K, Jung CW, Kim I, Yoon SS, Park S, Ahn JS, Yang DH, Lee JJ, Lee HS, Kim YS, Mun YC, Kim H, Park JH, Moon JH, Sohn SK, Lee SM, Lee WS, Kim KH, Won JH, Hyun MS, Park J, Lee JH, Shin HJ, Chung JS, Lee H, Eom HS, Lee GW, Cho YU, Jang S, Park CJ, Chi HS, Lee KH; Adult Acute Lymphoblastic Leukemia Working Party of the Korean Society of Hematology. Nilotinib combined with multiagent chemotherapy for newly diagnosed Philadelphia-positive acute lymphoblastic leukemia. Blood. 2015 Aug 6;126(6):746-56. doi: 10.1182/blood-2015-03-636548. Epub 2015 Jun 11. PMID 26065651
- [Background] Jain N, Maiti A, Ravandi F, Konopleva M, Daver N, Kadia T, Pemmaraju N, Short N, Kebriaei P, Ning J, Cortes J, Jabbour E, Kantarjian H. Inotuzumab ozogamicin with bosutinib for relapsed or refractory Philadelphia chromosome positive acute lymphoblastic leukemia or lymphoid blast phase of chronic myeloid leukemia. Am J Hematol. 2021 Aug 1;96(8):1000-1007. doi: 10.1002/ajh.26238. Epub 2021 May 28. PMID 33991360
- [Background] Vignetti M, Fazi P, Cimino G, Martinelli G, Di Raimondo F, Ferrara F, Meloni G, Ambrosetti A, Quarta G, Pagano L, Rege-Cambrin G, Elia L, Bertieri R, Annino L, Foa R, Baccarani M, Mandelli F. Imatinib plus steroids induces complete remissions and prolonged survival in elderly Philadelphia chromosome-positive patients with acute lymphoblastic leukemia without additional chemotherapy: results of the Gruppo Italiano Malattie Ematologiche dell'Adulto (GIMEMA) LAL0201-B protocol. Blood. 2007 May 1;109(9):3676-8. doi: 10.1182/blood-2006-10-052746. Epub 2007 Jan 9. PMID 17213285
- [Background] Rousselot P, Coude MM, Gokbuget N, Gambacorti Passerini C, Hayette S, Cayuela JM, Huguet F, Leguay T, Chevallier P, Salanoubat C, Bonmati C, Alexis M, Hunault M, Glaisner S, Agape P, Berthou C, Jourdan E, Fernandes J, Sutton L, Banos A, Reman O, Lioure B, Thomas X, Ifrah N, Lafage-Pochitaloff M, Bornand A, Morisset L, Robin V, Pfeifer H, Delannoy A, Ribera J, Bassan R, Delord M, Hoelzer D, Dombret H, Ottmann OG; European Working Group on Adult ALL (EWALL) group. Dasatinib and low-intensity chemotherapy in elderly patients with Philadelphia chromosome-positive ALL. Blood. 2016 Aug 11;128(6):774-82. doi: 10.1182/blood-2016-02-700153. Epub 2016 Apr 27. PMID 27121472
- [Background] Short NJ, Jabbour E, Sasaki K, Patel K, O'Brien SM, Cortes JE, Garris R, Issa GC, Garcia-Manero G, Luthra R, Thomas D, Kantarjian H, Ravandi F. Impact of complete molecular response on survival in patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Blood. 2016 Jul 28;128(4):504-7. doi: 10.1182/blood-2016-03-707562. Epub 2016 May 27. PMID 27235138
- [Background] Sasaki K, Kantarjian HM, Short NJ, Samra B, Khoury JD, Kanagal Shamanna R, Konopleva M, Jain N, DiNardo CD, Khouri R, Garcia-Manero G, Kadia TM, Wierda WG, Khouri IF, Kebriaei P, Mehta RS, Champlin RE, Garris R, Cheung CM, Daver N, Thompson PA, Yilmaz M, Ravandi F, Jabbour E. Prognostic factors for progression in patients with Philadelphia chromosome-positive acute lymphoblastic leukemia in complete molecular response within 3 months of therapy with tyrosine kinase inhibitors. Cancer. 2021 Aug 1;127(15):2648-2656. doi: 10.1002/cncr.33529. Epub 2021 Apr 1. PMID 33793964
- [Background] Short NJ, Kantarjian HM, Sasaki K, Ravandi F, Ko H, Cameron Yin C, Garcia-Manero G, Cortes JE, Garris R, O'Brien SM, Patel K, Khouri M, Thomas D, Jain N, Kadia TM, Daver NG, Benton CB, Issa GC, Konopleva M, Jabbour E. Poor outcomes associated with +der(22)t(9;22) and -9/9p in patients with Philadelphia chromosome-positive acute lymphoblastic leukemia receiving chemotherapy plus a tyrosine kinase inhibitor. Am J Hematol. 2017 Mar;92(3):238-243. doi: 10.1002/ajh.24625. Epub 2017 Feb 3. PMID 28006851
- [Background] Motllo C, Ribera JM, Morgades M, Granada I, Montesinos P, Mercadal S, Gonzalez-Campos J, Moreno MJ, Barba P, Cervera M, Barrios M, Novo A, Bernal T, Hernandez-Rivas JM, Abella E, Amigo ML, Tormo M, Martino R, Lavilla E, Bergua J, Serrano A, Garcia-Belmonte D, Guardia R, Grau J, Feliu E; PETHEMA Group, Spanish Society of Hematology. Frequency and prognostic significance of additional cytogenetic abnormalities to the Philadelphia chromosome in young and older adults with acute lymphoblastic leukemia. Leuk Lymphoma. 2018 Jan;59(1):146-154. doi: 10.1080/10428194.2017.1326596. Epub 2017 May 30. PMID 28554259
- [Background] Chiaretti S, Ansuinelli M, Vitale A, Elia L, Matarazzo M, Piciocchi A, Fazi P, Di Raimondo F, Santoro L, Fabbiano F, Califano C, Martinelli G, Ronco F, Ferrara F, Cascavilla N, Bigazzi C, Tedeschi A, Sica S, Di Renzo N, Melpignano A, Beltrami G, Vignetti M, Foa R. A multicenter total therapy strategy for de novo adult Philadelphia chromosome positive acute lymphoblastic leukemia patients: final results of the GIMEMA LAL1509 protocol. Haematologica. 2021 Jul 1;106(7):1828-1838. doi: 10.3324/haematol.2020.260935. PMID 33538150
- [Background] Short NJ, Kantarjian H, Jabbour E. SOHO State of the Art Updates & Next Questions: Intensive and Non-Intensive Approaches for Adults With Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia. Clin Lymphoma Myeloma Leuk. 2022 Feb;22(2):61-66. doi: 10.1016/j.clml.2021.08.003. Epub 2021 Aug 20. PMID 34561201
- [Background] Kim K, Jabbour E, Short NJ, Kebriaei P, Kantarjian H, Ravandi F. Current Approaches to Philadelphia Chromosome-Positive B-Cell Lineage Acute Lymphoblastic Leukemia: Role of Tyrosine Kinase Inhibitor and Stem Cell Transplant. Curr Oncol Rep. 2021 Jun 14;23(8):95. doi: 10.1007/s11912-021-01086-y. PMID 34125415
- [Background] Muffly L, Kebriaei P. Philadelphia chromosome positive acute lymphoblastic leukemia in adults: Therapeutic options and dilemmas in 2020. Semin Hematol. 2020 Jul;57(3):137-141. doi: 10.1053/j.seminhematol.2020.09.002. Epub 2020 Sep 11. PMID 33256903
- [Background] Ribera JM, Chiaretti S. Modern Management Options for Ph+ ALL. Cancers (Basel). 2022 Sep 20;14(19):4554. doi: 10.3390/cancers14194554. PMID 36230478
- [Background] Ansuinelli M, Cesini L, Chiaretti S, Foa R. Emerging tyrosine kinase inhibitors for the treatment of adult acute lymphoblastic leukemia. Expert Opin Emerg Drugs. 2021 Sep;26(3):281-294. doi: 10.1080/14728214.2021.1956462. Epub 2021 Jul 27. PMID 34259120
- [Background] Chiaretti S. Is Less More? Intensive Versus Non-Intensive Approach to Adults with Ph+ ALL. Clin Lymphoma Myeloma Leuk. 2020 Sep;20 Suppl 1:S54-S55. doi: 10.1016/S2152-2650(20)30461-4. No abstract available. PMID 32862869
- [Background] Ribera JM, Garcia O, Oriol A, Gil C, Montesinos P, Bernal T, Gonzalez-Campos J, Lavilla E, Ribera J, Brunet S, Martinez MP, Tormo M, Genesca E, Barba P, Sarra J, Monteserin MC, Soria B, Colorado M, Cladera A, Garcia-Guinon A, Calbacho M, Serrano A, Ortin X, Pedreno M, Amigo ML, Escoda L, Feliu E; PETHEMA Group, Spanish Society of Hematology. Feasibility and results of subtype-oriented protocols in older adults and fit elderly patients with acute lymphoblastic leukemia: Results of three prospective parallel trials from the PETHEMA group. Leuk Res. 2016 Feb;41:12-20. doi: 10.1016/j.leukres.2015.11.012. Epub 2015 Dec 2. PMID 26686475
- [Background] Ribera JM, Garcia-Calduch O, Ribera J, Montesinos P, Cano-Ferri I, Martinez P, Esteve J, Esteban D, Garcia-Fortes M, Alonso N, Gonzalez-Campos J, Bermudez A, Torrent A, Genesca E, Mercadal S, Martinez-Lopez J, Garcia-Sanz R. Ponatinib, chemotherapy, and transplant in adults with Philadelphia chromosome-positive acute lymphoblastic leukemia. Blood Adv. 2022 Sep 27;6(18):5395-5402. doi: 10.1182/bloodadvances.2022007764. PMID 35675590
- [Background] Giebel S, Marks DI, Boissel N, Baron F, Chiaretti S, Ciceri F, Cornelissen JJ, Doubek M, Esteve J, Fielding A, Foa R, Gorin NC, Gokbuget N, Hallbook H, Hoelzer D, Paravichnikova E, Ribera JM, Savani B, Rijneveld AW, Schmid C, Wartiovaara-Kautto U, Mohty M, Nagler A, Dombret H. Hematopoietic stem cell transplantation for adults with Philadelphia chromosome-negative acute lymphoblastic leukemia in first remission: a position statement of the European Working Group for Adult Acute Lymphoblastic Leukemia (EWALL) and the Acute Leukemia Working Party of the European Society for Blood and Marrow Transplantation (EBMT). Bone Marrow Transplant. 2019 Jun;54(6):798-809. doi: 10.1038/s41409-018-0373-4. Epub 2018 Nov 1. PMID 30385870
- [Background] Giebel S, Czyz A, Ottmann O, Baron F, Brissot E, Ciceri F, Cornelissen JJ, Esteve J, Gorin NC, Savani B, Schmid C, Mohty M, Nagler A. Use of tyrosine kinase inhibitors to prevent relapse after allogeneic hematopoietic stem cell transplantation for patients with Philadelphia chromosome-positive acute lymphoblastic leukemia: A position statement of the Acute Leukemia Working Party of the European Society for Blood and Marrow Transplantation. Cancer. 2016 Oct;122(19):2941-51. doi: 10.1002/cncr.30130. Epub 2016 Jun 16. PMID 27309127
- [Background] Saini N, Marin D, Ledesma C, Delgado R, Rondon G, Popat UR, Bashir Q, Hosing CM, Nieto Y, Alousi AM, Qazilbash MH, Ciurea S, Shpall E, Khouri I, Kantarjian H, Jabbour E, Ravandi F, Champlin RE, Kebriaei P. Impact of TKIs post-allogeneic hematopoietic cell transplantation in Philadelphia chromosome-positive ALL. Blood. 2020 Oct 8;136(15):1786-1789. doi: 10.1182/blood.2019004685. PMID 32492706
- [Background] Arber DA, Orazi A, Hasserjian RP, Borowitz MJ, Calvo KR, Kvasnicka HM, Wang SA, Bagg A, Barbui T, Branford S, Bueso-Ramos CE, Cortes JE, Dal Cin P, DiNardo CD, Dombret H, Duncavage EJ, Ebert BL, Estey EH, Facchetti F, Foucar K, Gangat N, Gianelli U, Godley LA, Gokbuget N, Gotlib J, Hellstrom-Lindberg E, Hobbs GS, Hoffman R, Jabbour EJ, Kiladjian JJ, Larson RA, Le Beau MM, Loh ML, Lowenberg B, Macintyre E, Malcovati L, Mullighan CG, Niemeyer C, Odenike OM, Ogawa S, Orfao A, Papaemmanuil E, Passamonti F, Porkka K, Pui CH, Radich JP, Reiter A, Rozman M, Rudelius M, Savona MR, Schiffer CA, Schmitt-Graeff A, Shimamura A, Sierra J, Stock WA, Stone RM, Tallman MS, Thiele J, Tien HF, Tzankov A, Vannucchi AM, Vyas P, Wei AH, Weinberg OK, Wierzbowska A, Cazzola M, Dohner H, Tefferi A. International Consensus Classification of Myeloid Neoplasms and Acute Leukemias: integrating morphologic, clinical, and genomic data. Blood. 2022 Sep 15;140(11):1200-1228. doi: 10.1182/blood.2022015850. PMID 35767897
- [Background] Lazaryan A, Dolan M, Zhang MJ, Wang HL, Kharfan-Dabaja MA, Marks DI, Bejanyan N, Copelan E, Majhail NS, Waller EK, Chao N, Prestidge T, Nishihori T, Kebriaei P, Inamoto Y, Hamilton B, Hashmi SK, Kamble RT, Bacher U, Hildebrandt GC, Stiff PJ, McGuirk J, Aldoss I, Beitinjaneh AM, Muffly L, Vij R, Olsson RF, Byrne M, Schultz KR, Aljurf M, Seftel M, Savoie ML, Savani BN, Verdonck LF, Cairo MS, Hossain N, Bhatt VR, Frangoul HA, Abdel-Azim H, Al Malki M, Munker R, Rizzieri D, Khera N, Nakamura R, Ringden O, Van der Poel M, Murthy HS, Liu H, Mori S, De Oliveira S, Bolanos-Meade J, Elsawy M, Barba P, Nathan S, George B, Pawarode A, Grunwald M, Agrawal V, Wang Y, Assal A, Caro PC, Kuwatsuka Y, Seo S, Ustun C, Politikos I, Lazarus HM, Saber W, Sandmaier BM, De Lima M, Litzow M, Bachanova V, Weisdorf D. Impact of cytogenetic abnormalities on outcomes of adult Philadelphia-negative acute lymphoblastic leukemia after allogeneic hematopoietic stem cell transplantation: a study by the Acute Leukemia Working Committee of the Center for International Blood and Marrow Transplant Research. Haematologica. 2021 Aug 1;106(8):2295-2296. doi: 10.3324/haematol.2021.279046. No abstract available. PMID 34333962
- [Background] Pfeifer H, Raum K, Markovic S, Nowak V, Fey S, Oblander J, Pressler J, Bohm V, Bruggemann M, Wunderle L, Huttmann A, Wasch R, Beck J, Stelljes M, Viardot A, Lang F, Hoelzer D, Hofmann WK, Serve H, Weiss C, Goekbuget N, Ottmann OG, Nowak D. Genomic CDKN2A/2B deletions in adult Ph+ ALL are adverse despite allogeneic stem cell transplantation. Blood. 2018 Mar 29;131(13):1464-1475. doi: 10.1182/blood-2017-07-796862. Epub 2018 Jan 18. PMID 29348129
- [Background] Paul S, Short NJ. Central Nervous System Involvement in Adults with Acute Leukemia: Diagnosis, Prevention, and Management. Curr Oncol Rep. 2022 Apr;24(4):427-436. doi: 10.1007/s11912-022-01220-4. Epub 2022 Feb 10. PMID 35141858
- See also: Web page of the sponsor of the study — http://www.fundacionpethema.es